CLINICAL TRIAL: NCT00958061
Title: CSP #579 - Long Term Health Outcomes of Women's Service During the Vietnam Era
Brief Title: Long Term Health Outcomes of Women Veterans' Service During the Vietnam Era
Acronym: Health ViEWS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 579
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Post-Traumatic Stress Disorder; Depression; Diabetes; Cardiovascular Disease
Keywords: CVD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vietnam-Era Women Veterans: For this study we will use a cohort of women who are on a roster of Vietnam Era women veterans (4,644 Vietnam, 1,213 near Vietnam, 5,465 non-Vietnam) previously identified and characterized by a review of their military personnel records and link it to a list of 8,061 women who presumably served in Southeast Asia. This final cohort could potentially contain approximately 14,000 women. After deceased individuals are removed from the active cohort and contact information is updated, we estimate that there could be approximately 10,000 women to whom the informed consent and mailed survey will be initially mailed.

SUMMARY:
Little is known about the long-term health and mental health status of women Vietnam veterans. For many of these women, the effects of this war are still present in their daily lives. As these women approach their mid-sixties, it is important to understand the impact of wartime deployment on health and mental health outcomes nearly 40 years later. The investigators propose to assess the prevalence of posttraumatic stress disorder (PTSD) and other mental and physical health conditions for women Vietnam veterans, and to explore the relationship between PTSD and other conditions and the Vietnam deployment experience. The investigators are interested in studying women Vietnam veterans who may have had direct exposure to traumatic events. For the first time, the investigators also want to study those who served in facilities near Vietnam. These women may have had similar, but less direct exposures. This cross-sectional study will seek to contact approximately 10,000 women for participation in a mailed survey, telephone interview and a review of their medical records. Women identified as serving in Vietnam, near Vietnam (in Asia during the Vietnam Ware) and in the U.S. during the Vietnam War will be identified from an established cohort and sent a survey on demographics, behaviors, disability, health-related quality of life, and medical conditions. Women agreeing to be contacted will also be interviewed by study investigators using the modified CIDI to ascertain current and lifetime mental health conditions (including PTSD) and exposure to traumatic events. A more extensive chart review will be conducted by a clinician to validate self-report of key medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women alive as of survey receipt who were active duty military personnel in one of the four Armed Services between July 4, 1965, and March 28, 1973, with a 30 day minimum period of service.
* This will include those who served in Vietnam, near Vietnam (Guam, the Philippines, Japan, Korea, Okinawa, or Thailand), or in the 50 United States.

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: For this study we will use a cohort of women who are on a roster of Vietnam Era women veterans (4,644 Vietnam, 1,213 near Vietnam, 5,465 non-Vietnam) previously identified and characterized by a review of their military personnel records and link it to a list of 8,061 women who presumably served in Southeast Asia. This final cohort could potentially contain approximately 14,000 women. After deceased individuals are removed from the active cohort and contact information is updated, we estimate that there could be approximately 10,000 women to whom the informed consent and mailed survey will be initially mailed.
Sampling Method: Probability Sample
Enrollment: 4219 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2012-08-07 (Actual); Study Completion 2012-08-07 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of lifetime and current psychiatric conditions including PTSD among women who served during the Vietnam Era. | two years
  The prevalence of lifetime and current psychiatric conditions including PTSD among women who served during the Vietnam Era.

SECONDARY OUTCOMES:
Characterize the physical health of women who served during the Vietnam Era. | two years
  Characterize the physical health of women who served during the Vietnam Era.
Characterize the level of current disability in women who served during the Vietnam Era. | two years
  Characterize the level of current disability in women who served during the Vietnam Era.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Magruder, PhD MPH BA, Study Chair — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kilbourne AM, Schumacher K, Frayne SM, Cypel Y, Barbaresso MM, Nord KM, Perzhinsky J, Lai Z, Prenovost K, Spiro A, Gleason TC, Kimerling R, Huang GD, Serpi TB, Magruder KM. Physical Health Conditions Among a Population-Based Cohort of Vietnam-Era Women Veterans: Agreement Between Self-Report and Medical Records. J Womens Health (Larchmt). 2017 Nov;26(11):1244-1251. doi: 10.1089/jwh.2016.6069. Epub 2017 Aug 7. PMID 28783423
- [Result] Schmidt EM, Magruder K, Kilbourne AM, Stock EM, Cypel Y, El Burai Felix S, Serpi T, Kimerling R, Cohen B, Spiro A, Furey J, Huang GD, Frayne SM. Four Decades after War: Incident Diabetes among Women Vietnam-Era Veterans in the HealthViEWS Study. Womens Health Issues. 2019 Nov-Dec;29(6):471-479. doi: 10.1016/j.whi.2019.08.002. Epub 2019 Sep 10. PMID 31519465
- [Result] Kimerling R, Serpi T, Weathers F, Kilbourne AM, Kang H, Collins JF, Cypel Y, Frayne SM, Furey J, Huang GD, Reinhard MJ, Spiro A, Magruder K. Diagnostic accuracy of the Composite International Diagnostic Interview (CIDI 3.0) PTSD module among female Vietnam-era veterans. J Trauma Stress. 2014 Apr;27(2):160-7. doi: 10.1002/jts.21905. PMID 24740869
- [Result] Kang HK, Cypel Y, Kilbourne AM, Magruder KM, Serpi T, Collins JF, Frayne SM, Furey J, Huang GD, Kimerling R, Reinhard MJ, Schumacher K, Spiro A 3rd. HealthViEWS: mortality study of female US Vietnam era veterans, 1965-2010. Am J Epidemiol. 2014 Mar 15;179(6):721-30. doi: 10.1093/aje/kwt319. Epub 2014 Jan 30. PMID 24488510
- [Result] Magruder K, Serpi T, Kimerling R, Kilbourne AM, Collins JF, Cypel Y, Frayne SM, Furey J, Huang GD, Gleason T, Reinhard MJ, Spiro A, Kang H. Prevalence of Posttraumatic Stress Disorder in Vietnam-Era Women Veterans: The Health of Vietnam-Era Women's Study (HealthVIEWS). JAMA Psychiatry. 2015 Nov;72(11):1127-34. doi: 10.1001/jamapsychiatry.2015.1786. PMID 26445103
- [Derived] Serier KN, Burns HM, Magruder KM, Spiro A, Pless Kaiser A, Kimerling R, Frayne SM, Kilbourne AM, Stock EM, Forsberg CW, Smith NL, Smith BN. Functioning and disability consequences of comorbid posttraumatic stress disorder and diabetes in Vietnam era men and women veterans. Health Psychol. 2025 Dec;44(12):1160-1170. doi: 10.1037/hea0001516. Epub 2025 Jun 12. PMID 40504650